CLINICAL TRIAL: NCT04860167
Title: Propofol Sedation During Endoscopic Retrograde Cholangiopancreatography: A Comparison Between Conventional Versus Bispectral Index Guided Approach and Effect of Diclofenac Sodium Along With Topical Pharyngeal Anaesthesia
Brief Title: Sedation for Patients Undergoing Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Gaurav Sindwani, Associate professor, Department of Anaesthesiology, Principal Investigator, Institute of Liver and Biliary Sciences, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBSIndia3
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Biliary Colic
Keywords: Diclofenac; Propofol; Topical anaesthesia
MeSH Terms: interventions — Propofol; Diclofenac; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (No Intervention): The intravenous infusion of propofol was administered for ERCP procedure based on clinical judgment and the patient's requirement.
- Group B (Active Comparator): The intravenous infusion of propofol was administered for ERCP procedure titrated to BIS value 60-80.
  Interventions: Drug: Propofol
- Group C (Active Comparator): Patients received 75 mg of inj. Diclofenac sodium (diluted in 100 ml of 0.9 % normal saline) intravenously 30 mins before the start of procedure & topical pharyngeal anesthesia with 4 squirts of 10% lidocaine spray ( one squirt each to posterior pharyngeal wall, base of tongue, and bilateral palatoglossal and palatopharyngeal folds ) 5 mins before the start of ERCP procedure. Intravenous infusion of propofol was administered for ERCP procedure titrated to BIS value 60-80.
  Interventions: Drug: Diclofenac Sodium and Lignocaine 10 % spray

INTERVENTIONS:
Drug: Propofol — Injection propofol was given to keep the BIS value 60-80 during the ERCP procedure
  Other Names: Neorof
  Arms: Group B
Drug: Diclofenac Sodium and Lignocaine 10 % spray — Injection Diclofenac sodium was given in the preoperative area 30 minutes before the procedure and four squirts of 10% lignocaine were given 5 minutes prior to the start of the procedure
  Other Names: Dynapar
  Arms: Group C

SUMMARY:
This study was performed to evaluate the role of BIS monitored sedation in reducing the dose of propofol and to know the effectiveness of pre-procedure administration of intravenous diclofenac sodium along with topical pharyngeal anesthesia in reducing the dose of propofol in patients undergoing endoscopic retrograde cholangiopancreatography.

DETAILED DESCRIPTION:
It was a single-center open-labeled Prospective Randomized study. After approval of the study by the institutional ethical committee & obtaining written informed consent, 90 patients scheduled for ERCP procedure were randomized by using the block randomization method into the following three groups, Group A (n=30)-The intravenous infusion of propofol was administered for the ERCP procedure based on clinical judgment and the patient's requirement.

Group B (n=30) - The intravenous infusion of propofol was administered for ERCP procedure titrated to BIS value 60-80.

Group C (n=30) - Patients received 75 mg of inj. Diclofenac sodium (diluted in 100 ml of 0.9 % normal saline) intravenously 30 mins before the start of procedure & topical pharyngeal anesthesia with 4 squirts of 10% lidocaine spray ( one squirt each to posterior pharyngeal wall, base of tongue, and bilateral palatoglossal and palatopharyngeal folds ) 5 mins before the start of ERCP procedure. Intravenous infusion of propofol was administered for ERCP procedure titrated to BIS value 60-80.

In all three groups, after completing the standard pre-anesthesia checklist, patients were positioned in the semi prone-position and standard ASA monitors were attached (electrocardiogram, pulse oximetry, and non-invasive blood pressure, EtCO2). Also, the BIS monitor was attached in group B & group C. Baseline values were noted before the start of sedation. Supplemental oxygen was provided by nasal prongs @ 2/min. Patients in all groups were sedated with an initial bolus dose of fentanyl 1 mcg/kg & propofol 1-1.5 mg/kg intravenously. Sedation was maintained with propofol infusion at the rate of 80-100 mcg/kg/min. In group A, propofol sedation was further titrated based on clinical judgment and patient's requirement. Whereas in group B & group C, propofol sedation was further titrated to maintain a BIS value between 60-80. If the patient moves despite BIS 60-80, an additional bolus of 30 mg i.v. propofol was administered. In addition to these, i.v. fentanyl 25mcg was administered as a rescue analgesic.All pre-procedure drugs were administered in the preoperative room with standard ASA monitoring.

Hemodynamic parameters were monitored at 5-min intervals. The incidence and number of episodes of patient's movements, cough/gag reflex, and hiccups were noted. The incidence of desaturation (fall in oxygen saturation < 94 % with oxygen supplementation), hypotension (17) (defined as systolic blood pressure < 90 mm of Hg ), and bradycardia (defined as HR < 50 beats per minute) was also be noted. Standard anesthesia protocol was followed for the management of desaturation and hemodynamic instability. Desaturation was managed by chin lift & jaw thrust maneuver. The nasal airway was inserted if deemed necessary by the concerned anesthetist. Further, if desaturation persists & lack of respiratory effort is seen for more than 20 seconds, sedation was discontinued, and mask ventilation is initiated in the lateral position. Insertion of supraglottic airway devise or tracheal intubation (after turning the patient supine) performed as per anesthetist discretion and the patient will be excluded from the study. Hypotension managed with 6-12 mg of intravenous ephedrine or a fluid bolus of 500 cc of plasmalyte. Bradycardia is managed by 0.6 mg of intravenous atropine.

At the end of the procedure, propofol infusion was stopped and the total dose of propofol administered in mg/kg/hr was calculated. Thereafter, time to achieve eye-opening to verbal commands was calculated.

Post-procedure, patients were nursed in the left lateral position, and vitals (HR, NIBP, SpO2) was noted every 5 mins. Also, readiness to discharge is assessed by the noting post-anesthesia discharge score (PADS) every 15 mins. For patients having breakthrough pain, 1 gram iv paracetamol was administered in all the groups. The endpoint of complete recovery was a PADS score of 10. Also at the end of the procedure, the endoscopist was asked to grade ease of procedure based on 1=poor, 2=fair, 3=acceptable, 4=good, 5=excellent scale.

At the time of discharge, the patient's satisfaction for the ERCP procedure was grade on 1=unacceptable, 2=extremely uncomfortable, 3=slightly uncomfortable, 4=no discomfort scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 yrs
2. ASA I & II

Exclusion Criteria:

1. Age < 18 yrs & > 65 yrs
2. ASA III & IV patients
3. Chronic Liver Disease
4. Pregnant patients
5. Patients with a history of (H/O) Drug abuse
6. Patients refusing consent
7. H/o Acute kidney injury
8. H/o allergy to propofol / lidocaine/ NSAIDS
9. Post liver transplant patients
10. Patients with h/o egg allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Total dose of propofol required in mg/kg/hr during ERCP procedure among different groups. | 2 hours
  Total dose of propofol required to complete the ERCP procedure was noted

SECONDARY OUTCOMES:
Mean recovery time between different groups. | 24 hours
  Total time taken by the patient to reach a post-anesthesia discharge score of 10 was taken as the mean recovery time
Time taken to achieve eye opening to verbal stimulus among different groups | 24 hours
  Total time taken by the patient to open eyes in response to the verbal commands after the propofol was stopped
Incidence of hypotension, bradycardia, limb movements and gag reflex during the ERCP procedure | 24 hours
  Incidence of hypotension, bradycardia, limb movement and gag reflex was noted during the ERCP procedure

CONTACTS AND LOCATIONS:
Overall Officials: gaurav sindwani, md, Principal Investigator — ilbs
Locations (1):
- Gaurav Sindwani, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patai A, Solymosi N, Mohacsi L, Patai AV. Indomethacin and diclofenac in the prevention of post-ERCP pancreatitis: a systematic review and meta-analysis of prospective controlled trials. Gastrointest Endosc. 2017 Jun;85(6):1144-1156.e1. doi: 10.1016/j.gie.2017.01.033. Epub 2017 Feb 4. PMID 28167118
- [Result] Quesada N, Judez D, Martinez Ubieto J, Pascual A, Chacon E, De Pablo F, Minchole E, Bello S. Bispectral Index Monitoring Reduces the Dosage of Propofol and Adverse Events in Sedation for Endobronchial Ultrasound. Respiration. 2016;92(3):166-75. doi: 10.1159/000448433. Epub 2016 Sep 7. PMID 27598398
- [Result] Wehrmann T, Grotkamp J, Stergiou N, Riphaus A, Kluge A, Lembcke B, Schultz A. Electroencephalogram monitoring facilitates sedation with propofol for routine ERCP: a randomized, controlled trial. Gastrointest Endosc. 2002 Dec;56(6):817-24. doi: 10.1067/mge.2002.129603. PMID 12447291
- [Result] White PF, Sacan O, Tufanogullari B, Eng M, Nuangchamnong N, Ogunnaike B. Effect of short-term postoperative celecoxib administration on patient outcome after outpatient laparoscopic surgery. Can J Anaesth. 2007 May;54(5):342-8. doi: 10.1007/BF03022655. PMID 17470884
- [Result] Paspatis GA, Chainaki I, Manolaraki MM, Vardas E, Theodoropoulou A, Tribonias G, Konstantinidis K, Karmiris K, Chlouverakis G. Efficacy of bispectral index monitoring as an adjunct to propofol deep sedation for ERCP: a randomized controlled trial. Endoscopy. 2009 Dec;41(12):1046-51. doi: 10.1055/s-0029-1215342. Epub 2009 Dec 4. PMID 19967620